CLINICAL TRIAL: NCT03823768
Title: The Effect of Conversion to Once-Daily Envarsus® on the Neurologic Toxicity Burden in Liver Transplant Recipients
Brief Title: Envarsus Neurotoxicity Burden in Liver Transplant Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Veloxis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, David J. Taber, Professor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00083855
Record Dates: First submitted 2019-01-29; First posted 2019-01-30 (Actual); Results first posted 2024-06-27 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Neurotoxicity; Liver Transplant; Complications
MeSH Terms: conditions — Neurotoxicity Syndromes | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm 1: Control (Active Comparator): Tacrolimus immediate release twice daily for 6 months
  Interventions: Drug: Tacrolimus Immediate release
- Arm 2: Intervention (Experimental): Envarsus daily for 6 months.
  Interventions: Drug: Envarsus

INTERVENTIONS:
Drug: Envarsus — Subjects in this group will take Envarsus daily for 6 months of treatment (goal 24 hour trough: 3-10 ng/mL) +/- adjunctive agent and prednisone.
  Arms: Arm 2: Intervention
Drug: Tacrolimus Immediate release — Subjects in this group will take Tacrolimus immediate release for 6 months of treatment (goal 12 hour trough: 3-10 ng/mL) +/- adjunctive agent and prednisone.
  Arms: Arm 1: Control

SUMMARY:
This study will compare neurologic side effects associated with two immunosuppressant medications used in liver transplant patients. The standard therapy of twice daily immediate release Tacrolimus will be compared to Envarsus once daily. We hypothesize that Envarsus will show a lower rate of neurologic side effects than immediate release tacrolimus.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adult (≥18 years old) with a history of liver or liver/kidney transplant within the first 6 months of transplant.
2. Patients must be capable of understanding the purposes and risks of the study and have the ability to give written informed consent and be willing to participate and comply with the study.

Exclusion Criteria:

1. Patients will be excluded if they are pregnant or nursing females or males with a pregnant female partner
2. HIV positive (HIV ab +)
3. Unable to tolerate oral medications
4. Use of another investigational product within thirty days prior to receiving study medication
5. Moderate acute cellular rejection (RAI ≥ 5) within the past month
6. A condition that is known to cause tremor such as essential tremor, Parkinson disease, or enhanced physiologic tremor.
7. Patients taking medications known to induce tremors or dopamine blocking agents
8. A condition or disorder that, in the opinion of the investigator, may adversely affect the outcome of the study or the safety of the subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2024-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Derek Dubay, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Derived] Coffman KS, Revuelta GJ, DeTurk N, Palmer C, Culpepper H, Overstreet M, Fleming J, Terry K, Patel N, McGillicuddy J, Nagaraju S, Rice TC, Taber DJ. Results of a Randomized Controlled Trial Evaluating the Impact of Conversion to LCP Tacrolimus on Neurologic Toxicities in Liver Transplant Recipients. Int J Hepatol. 2025 Oct 6;2025:4374144. doi: 10.1155/ijh/4374144. eCollection 2025. PMID 41089174

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1: Control | Arm 2: Intervention
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Control | Arm 2: Intervention | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 14 | 28
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (13) | 52 (9) | 52 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 13 | 22
  Male | 6 | 2 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 14 | 13 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in Neurotoxicity Burden
Description: Estimate the change from baseline to six months in neurotoxicity burden measured by a composite Patient Global Impression of Improvement score (PGI-I, with a range of 4-28) The PGI-I is a global index that may be used to rate the response of a condition to a therapy (transition scale). Scale min=4, scale max=28. The scale is made up of four questions, each question has a total of 7 responses, the total score is the sum of each questions choice (1-7). Higher values represent a worsening condition. A score of 16 would indicate no overall change. A score of 15 or lower indicates improvement in the condition and a score of 17 or higher indicates a worsening of the condition. A score of 28 would indicate "very much worse," while a score of 4 would indicate "very much better." A relative change of 2 points would be considered a significant change from baseline.
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm 1: Control | Arm 2: Intervention
Number analyzed (Participants) | 15 | 15
score on a scale | -5 [-13.5 to -0.25] | -4 [-9.5 to -0.5]

ADVERSE EVENTS:
Time Frame: 6 months post-transplant
Description: SAE was defined as a hospitalization, prolonged hospitalization, graft loss or death.
Arm/Group | Arm 1: Control | Arm 2: Intervention
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 1/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Control (N=15) | Arm 2: Intervention (N=15)
Acute Rejection (Gastrointestinal disorders) | 0 (0) | 1 (1) — Liver rejection

LIMITATIONS AND CAVEATS:
Study conducted during COVID 19 pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-10): https://cdn.clinicaltrials.gov/large-docs/68/NCT03823768/Prot_SAP_000.pdf